CLINICAL TRIAL: NCT03741803
Title: Randomized Controlled Trial to Evaluate the Relationship Between Delayed Cord Clamping at Birth and Neonatal Bilirubin Levels in Parturients With a Prior Child Requiring Therapy for Neonatal Jaundice
Brief Title: Relationship Between Delayed Cord Clamping at Birth and Neonatal Bilirubin Levels in Parturients With a Prior Child Requiring Therapy for Neonatal Jaundice
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Study paused due to COVID-19 and personnel
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Pamela Berens, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-MS-17-0803
Record Dates: First submitted 2018-11-12; First posted 2018-11-15 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Hyperbilirubinemia, Neonatal; Jaundice, Neonatal
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal; Jaundice, Neonatal | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Delayed cord clamping (Active Comparator)
  Interventions: Procedure: Delayed cord clamping
- Early cord clamping (Active Comparator)
  Interventions: Procedure: Early cord clamping

INTERVENTIONS:
Procedure: Delayed cord clamping — The umbilical cord will be clamped after 60 seconds after birth
  Arms: Delayed cord clamping
Procedure: Early cord clamping — The umbilical cord will be clamped as soon as feasible after birth, usually within the initial 15 seconds after birth.
  Arms: Early cord clamping

SUMMARY:
The purpose of the study is to determine if neonates (who already have an increased risk of hyperbilirubinemia due to mother's history of having previous neonate who received phototherapy for hyperbilirubinemia) have higher bilirubin levels 24 hours after birth with delayed cord clamping.

ELIGIBILITY:
Inclusion Criteria:

* mothers delivering at 35 weeks or greater
* mothers who have had at least 1 previous child that received phototherapy for hyperbilirubinemia
* multiple gestations can be included unless the neonate does not meet criteria for delayed cord clamping as described below or due to concerns about safety of delayed cord clamping for timing of delivery of the 2nd twin (ie: 2nd twin requires immediate delivery intervention)

Exclusion Criteria:

- Neonates who do not meet criteria for delayed cord clamping (any infant that any provider in the room felt needed evaluation by the neonatal transport team immediately so that the infant would be handed off for resuscitation. If the patient required delivery by cesarean section the delayed cord clamping protocol would be abandoned).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-11-09 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Neonatal bilirubin level | 24 hours after birth

SECONDARY OUTCOMES:
Number of neonates with hyperbilirubinemia | 24 hours after birth
  Hyperbilirubinemia is a condition in which there is too much bilirubin in the blood.
Number of neonates with a need for phototherapy | From birth to up to 1 week after birth
Number of neonates with a need for exchange transfusion | From birth to up to 1 week after birth
Number of neonates admitted to the neonatal intensive care unit (NICU) | From birth to up to 1 week after birth
Number of mothers with postpartum hemorrhage | From birth to up to 1 week after birth
Number of neonates re-hospitalized for jaundice | From birth to up to 1 week after birth

CONTACTS AND LOCATIONS:
Overall Officials: Pamela D Berens, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No